CLINICAL TRIAL: NCT05930847
Title: Effect of Respiratory Training Digital Game on Respiratory Functions, and Psychological Status in Childhood Asthma
Brief Title: Digital Respiratory Game in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozden Gokcek, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/16
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Asthma in Children
Keywords: Digital game; Pediatric asthma; Quality of life; Respiratory training; Psychological status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital game group (Experimental): In addition to routine drug use, children of the digital game group were followed up with 15 sessions of 15 minutes of digital games for respiratory training.
  Interventions: Device: Digital Game Application; Drug: Use of medication for asthma
- Routine medical treatment group (Active Comparator): The children continued their current asthma treatment in the same way. They did not receive any extra treatment.
  Interventions: Drug: Use of medication for asthma

INTERVENTIONS:
Device: Digital Game Application — The digital game contains brief information about the respiratory system adapted to children, and it is a game whose duration can be adjusted manually to follow the treatment process of the patient, taking into account the ½ ratio in the inhalation and exhalation process in the clinic.
  Arms: Digital game group
Drug: Use of medication for asthma — The children continued to take their current asthma medication on the same schedule. The drugs used by the children were zespira and ventolin.

SUMMARY:
This study aims to examine the effects of a digital game designed for respiratory training in childhood asthma. Fifteen children aged 8-14 years with asthma were included in the study. There were two groups a digital game group (n=9) and a control group (n=6). Respiratory training was given to the digital game group with a digital game. The control group was followed with medication. Both groups were evaluated at baseline and after 3 weeks.

DETAILED DESCRIPTION:
Asthma is a chronic obstructive disease that is common in children worldwide. This study aims to examine the effects of a digital game designed for respiratory training in childhood asthma.

Fifteen children aged 8-14 years with asthma were included in the study. There were two groups a digital game group (n=9) and a control group (n=6). Demographic information of the children was recorded. Pulmonary function test (PFT) was evaluated with a portable spirometer (Spirobank MIR), the quality of life of the children was evaluated with the Paediatric Asthma Quality of Life Questionnaire and psychological status was evaluated with the child depression scale. Respiratory training was given to the digital game group with a digital game. The control group was followed with medication. Both groups were evaluated at baseline and after 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with asthma according to GINA criteria
* Cooperative

Exclusion Criteria:

* Presence of neurological problems
* Presence of systemic disorders

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test (PFT) | 6 months
  The respiratory function of the children was evaluated with a portable spirometer (Spirobank MIR, Italy) according to the European Respiratory Society (ERS) and American Thoracic Society (ATS) criteria. The test will be performed in a sitting position, with the patient asked to inhale deeply and then exhale rapidly through the spirometer.

SECONDARY OUTCOMES:
The Pediatric Asthma Quality of Life Questionnaire (PAQLQ) | 6 months
  It is used to evaluate the quality of life of children aged 7-17 years by measuring the physical, mental, and social impairment specific to asthma. It is a 23-item quality-of-life scale developed to measure the physical, mental, and social disorders of children with asthma. The total score for all items is 23-161. Higher scores suggest a better quality of life.
Childhood Depression Inventory (CDI) | 4 months
  The depression status of the children was evaluated with the Child Depression Scale. In this 27-item scale, 1,2,3 items are specified for each question and the scoring is done on a maximum of 54 points, with 0 for 1, 1 for 2 and 2 for 3. The cut-off score is recommended as 19 and the severity of depression increases as the score increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university faculty of health sciences, Izmir, Karsıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data sets generated and/or analyzed during the current study are available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP